CLINICAL TRIAL: NCT05211674
Title: Quantified Analysis of Postural Control of COPD Patients During Tasks of Daily Living
Brief Title: Analysis of Postural Control of COPD Patients (ATTRACTION)
Acronym: ATTRACTION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Rennes 2 (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Principal Investigator, Graziella Brinchault, Principal investigator, Rennes University Hospital
Other Study IDs: M2S-ATTRACTION
Record Dates: First submitted 2021-11-23; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; postural balance; activities of daily living
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients
  Interventions: Other: quantified analysis of postural control during activities of daily living
- Healthy controls
  Interventions: Other: quantified analysis of postural control during activities of daily living

INTERVENTIONS:
Other: quantified analysis of postural control during activities of daily living — functional tests that reproduce tasks of daily living (timed up and go test with and without dual cognitive task, modified Glittre ADL test)

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common chronic respiratory disease, causing disabling respiratory symptoms and impairing patients' quality of life. Currently one of the leading causes of death worldwide, COPD is a major socio-economic concern. It is also accompanied by extremely frequent extra-respiratory manifestations (or co-morbidities). Among these secondary manifestations, the equilibrium of these patients is subject to modifications: thus, numerous studies have shown that the equilibrium of COPD patients was altered compared to healthy age-matched subjects. This alteration is associated with a greater functional limitation and a higher risk of falling. Although this impairment has been demonstrated clinically, the balance of these patients has never been analysed using quantified movement analysis tools during tasks similar to those performed in daily life. Moreover, the underlying mechanisms remain unknown and the possible associations with several clinical factors of interest (pain, dyspnea, muscle function...) have not yet been assessed. The hypotheses of this project are that (1) the postural control of COPD patients is altered compared to healthy subjects during tasks of daily living and these changes can be characterised. (2) Several clinical factors are associated with these changes.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients GOLD stage 2 and 3 (A-D)
* In accordance with Article L1121-8-1 of the Public Health Code, participants must be affiliated to a social security scheme or benefit from such a scheme.

Exclusion Criteria:

1. the presence of long-term or exercise-based oxygen therapy,
2. the presence of a medically diagnosed pathology causing manifest disorders of balance,
3. the inability to walk 150 m without stopping and to climb or descend stairs,
4. a history of pneumonectomy or lobectomy within the last six months,
5. the existence of an acute respiratory exacerbation within the last two months,
6. the presence of obvious cognitive impairment that impairs comprehension of instructions,
7. body mass index less than 21 or more than 35 kg/m².
8. Person referred to in articles L. 1121-5 to L. 1121-8 and L. 1121-12 of the public health code:

   * Pregnant woman, woman in labour or nursing mother
   * Person deprived of liberty by judicial or administrative decision
   * Person hospitalised without consent and not subject to a legal protection measure, and person admitted to a health or social establishment for purposes other than research
   * Minor
   * Person subject to a period of exclusion for other research
   * Person of full age subject to a legal protection measure (guardianship, curatorship or safeguard of justice), person of full age unable to express their consent and not subject to a protection measure
9. Person under psychiatric care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients that realize their medical follow-up at University Hospital of Rennes
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Margins of stability | Clinical assessment at baseline
  Postural control parameter related to the centre of mass (CoM) and the base of support of the participant, assessed during the functional tests
Margins of stability variability | Clinical assessment at baseline
  Coefficient of variation of a postural control parameter related to the centre of mass (CoM) and the base of support of the participant, assessed during the functional tests
Center of Mass velocity | Clinical assessment at baseline
  Parameter of participant's Centre of Mass (CoM) during the functional tests
Center of mass displacement | Clinical assessment at baseline
  Parameter of participant's Centre of Mass (CoM) during the functional tests

SECONDARY OUTCOMES:
Evolution of articular angulations | Clinical assessment at baseline
  Articular angulations assessed at the ankle, knee, hip, spine and thoracic level during the functional tests
Centre of pressure (CoP) Area | Clinical assessment at baseline
  Parameter of participant's Centre of Pressure (CoP) during the sit to stand and stand to sit tasks of the Glittre-ADL test
Centre of pressure (CoP) velocity | Clinical assessment at baseline
  Parameter of participant's Centre of Pressure (CoP) during the sit to stand and stand to sit tasks of the Glittre-ADL test
Centre of pressure (CoP) variability | Clinical assessment at baseline
  Coefficient of variation of participant's Centre of Pressure (CoP) during the sit to stand and stand to sit tasks of the Glittre-ADL test
Gait Cadence | Clinical assessment at baseline
  spatio-temporal parameter of gait assessed during the walking part of the Glittre-ADL test
Gait velocity | Clinical assessment at baseline
  spatio-temporal parameter of gait assessed during the walking part of the Glittre-ADL test
Gait phases duration | Clinical assessment at baseline
  spatio-temporal parameter of gait assessed during the walking part of the Glittre-ADL test
Step width | Clinical assessment at baseline
  spatio-temporal parameter of gait assessed during the walking part of the Glittre-ADL test
Step length | Clinical assessment at baseline
  spatio-temporal parameter of gait assessed during the walking part of the Glittre-ADL test
Completion time of the Modified Glittre ADL | Clinical assessment at baseline
  Time to complete the modified Glittre-ADL test
Completion time of the timed up and go test | Clinical assessment at baseline
  Time to complete the timed up and go test test

OTHER OUTCOMES:
Dyspnea assessment scale | Clinical assessment at baseline
  assessed by the modified Borg Scale which is a 0 to 10 scale (0 representing no dyspnea, 10 representing the worst imaginable dyspnea). Dyspnea is assessed before, during and after the functional tests
Heart rate | Clinical assessment at baseline
  assessed before, during and after functional tests
Leg discomfort scale | Clinical assessment at baseline
  assessed on a 0 to 10 scale (0 representing no discomfort, 10 representing the worst imaginable discomfort).Leg discomfort is assessed before, during and after the functional tests
Visual analog scale for pain | Clinical assessment at baseline
  Pain is assessed by a visual analog scale which is a 100mm long horizontal line with verbal descriptors at each end to express the extremes of the feeling (Here no pain and the worst imaginable pain)
Pain Drawing scale | Clinical assessment at baseline
  participants are invited to identify on a body chart the location of experienced pain.
Multi-dimensional dyspnea profile (MDP) | Clinical assessment at baseline
  Dyspnea assessment tool which investigates sensory and affective dimensions of dyspnea
London chest activity of daily living questionnaire (LCADL) | Clinical assessment at baseline
  Dyspnea assessment tool which investigates the impact of dyspnea on 15 activities of daily living. A score from 0 to 5 is given for each activity, 5 representing an higher impact of dyspnea on the activity.
Modified Medical Research Council Scale (MMRC) | Clinical assessment at baseline
  Dyspnea assessment tool which investigates impact of dyspnea in participants life. This is a 0 to 4 scale with descriptors associated to each number. 4 representing the most severe impact of dyspnea.
Charlson Index | Clinical assessment at baseline
  Comorbidities assessment tool which list 19 potential comorbidities associated with a weighted score. The points are attributed when the comorbidity is present. A total score is then calculated. An higher score indicates an higher severity.
Body composition | Clinical assessment at baseline
  Determination of fat free mass and fat mass by bioelectrical impedance analysis.
Maximal inspiratory pressure | Clinical assessment at baseline
  inspiratory muscles strength assessment
Falls Efficacy Scale - International | Clinical assessment at baseline
  Fear of falling assessment tool which investigates fear of falling in 16 different activities. Each activity is scored from 0 to 4 (4 representing an higher fear of falling in this activity). The total score range from 16 to 64 (an higher score indicating a most severe fear of falling)
Number of anterior falls | Clinical assessment at baseline
  assessment of fall occurence in the last 12 months
General Practioner assessment of Cognition (GP-COG) | Clinical assessment at baseline
  assessment of cognitive function. GP-COG gives a score from 0 to 9 (9 indicating a better cognitive function)
International Physical Activity Questionnaire (IPAQ short-form) | Clinical assessment at baseline
  assessment of daily physical activity and sedentarity
COPD assessment test (CAT) | Clinical assessment at baseline
  quality of life assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Brinchault, MD, Principal Investigator — University Hospital of Rennes

IPD SHARING:
Plan to Share IPD: Undecided